CLINICAL TRIAL: NCT06245343
Title: Investigation of the Effects of Functional Inspiratory Muscle Training on Oxygen Consumption, Muscle Oxygenation, Balance and Physical Activity Level in Patients With Lung Cancer
Brief Title: Investigation of the Effects of Functional Inspiratory Muscle Training in Patients With Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Study director, PT, PhD, Prof. Dr. Faculty of Health Sciences, Department of Cardiopulmonary Physiotherapy and Rehabilitation, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Gazi University 80
Record Dates: First submitted 2024-01-21; First posted 2024-02-07 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Oxygen consumption; Muscle oxygenation; Balance; Physical activity; Functional inspiratory muscle training
MeSH Terms: conditions — Lung Neoplasms; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple-blind study; the patients will not be informed about training group or control group and they will be evaluated and trained at different places and times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional inspiratory muscle training group (Experimental): Patients in the training group will be performed functional inspiratory muscle training with the PowerBreathe® (inspiratory muscle training device) device at 50% of the maximal inspiratory pressure.
  Interventions: Device: Functional inspiratory muscle training group
- Control group (Sham Comparator): The control group will not be given any training during the study period.
  Interventions: Device: Control group

INTERVENTIONS:
Device: Functional inspiratory muscle training group — Patients will be given fundamental inspiratory muscle training with the inspiratory muscle training device at 50% of the maximal inspiratory pressure 30 min/day, 3 days/week for 4 weeks online with a physiotherapist. On the other days of the week, the training will be used as a home program.
  In the 5th week, the functional inspiratory muscle training program will be started. Before the program begins, patients will be shown the exercises in the functional inspiratory muscle training program. Patients will be given functional inspiratory muscle training with the inspiratory muscle training device at 50% of the maximal inspiratory pressure 30 min/day, 3 days/week for 4 weeks online with a physiotherapist. On the other days of the week, fundamental inspiratory muscle training will be used as a home program.
  Pressure increases will be made weekly to 10 centimeters of water (cmH2O). Unsupervised training sessions will be followed by charts filled out by patients.
  Arms: Functional inspiratory muscle training group
Device: Control group — The control group will not be given any training during the 8-week period. After the study, the treatment applied to the training group will also be applied to the control group in order to ensure that the patients in the control group are not ethically deprived of rehabilitation.
  Arms: Control group

SUMMARY:
Patients' pulmonary functions and diffusion capacity worsen following lung cancer surgery. Diaphragmatic activity and lung compliance decrease due to surgery. Peripheral and respiratory muscle functions are impaired in patients with lung cancer, exercise capacity and physical activity level decreased. Patients have postural instability and balance problems. Inspiratory muscle training has increased inspiratory muscle strength in patients with lung cancer. However, there is no study investigating functional inspiratory muscle training in patients with lung cancer.

DETAILED DESCRIPTION:
Lung cancer is a malignant lung tumor characterized by uncontrolled cell growth in lung tissues. The main treatment methods for lung cancer are chemotherapy, radiotherapy, and surgery. Molecularly targeted therapy and immunotherapy are also among the treatment options. Patients with lung cancer experience various symptoms such as dyspnea, cough, chest pain, hemoptysis, fatigue, weight loss due to the disease process, the effects of chemotherapy and radiotherapy treatment, and comorbidities. The treatment method varies depending on the histological type, stage, location of the tumor, and the physical condition of the patient. Surgery is performed as a therapeutic option for many patients with lung cancer. Lung cancer surgery impair the cardiorespiratory functions of the patients. Patients' pulmonary functions and diffusion capacity worsen following lung cancer surgery. In lung cancer patients, the incision applied to the respiratory muscles due to surgery and changes in the mechanics of the chest wall cause worsening of respiratory muscle function. The condition results in dyspnea in patients at rest and during activities of daily living. Mitochondrial dysfunction due to the pathogenesis of the disease and chemotherapy/radiotherapy leads to deterioration in muscle oxygen metabolism. In individuals with reduced muscle oxygen, exercise tolerance and muscle strength decrease. Impairment of diaphragm function is associated with decreased postural stability after lung cancer surgery. Patients with lung cancer have postural instability and balance problems. Lung cancer significantly affects the quality of life of patients, limiting their physical and social activities. Inspiratory muscle training is recommended as part of disease management for lung cancer. In the literature, there are studies investigating the effectiveness of inspiratory muscle training in lung cancer patients in the preoperative, perioperative, and postoperative periods. However, there is no study investigating functional inspiratory muscle training in patients with lung cancer. Functional inspiratory muscle training (IMT) was developed by McConnell. It is a program that is based on the functions of respiratory muscles other than breathing, and IMT is applied along with exercise.

The primary aim of this study: To investigate the effects of functional inspiratory muscle training on oxygen consumption, muscle oxygenation, balance and physical activity level in patients with lung cancer.

The secondary aim of this study: To investigate the effects of functional inspiratory muscle training on pulmonary functions, peripheral and respiratory muscle strength, inspiratory and trunk muscle endurance, cough strength, fatigue, dyspnea and quality of life in patients with lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-80 years with lung cancer
2. Patients who have undergone surgical treatment (wedge resection, segmentectomy, lobectomy, bilobectomy) for lung cancer
3. Lung cancer treatment completed, in remission and under follow-up

Exclusion Criteria:

1. According to the American Association of Sports Medicine (ACSM) with absolute and relative contraindications to exercise tests
2. Patients who are having comorbidities such as uncontrolled hypertension, diabetes mellitus, heart failure or atrial fibrillation
3. Patients who are having acute infection during evaluation
4. Patients who are having orthopedic, neurological, psychological, etc. problems that limit evaluations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Oxygen Consumption | Trough study completion, an average of 2 year
  Maximum exercise capacity will be assessed by symptom-limited cardiopulmonary exercise testing on a treadmill at gradually increasing speed and degree, and oxygen consumption will be measured during the test.
Muscle oxygenation | Trough study completion, an average of 2 year
  Muscle oxygenation of the quadriceps femoris (during the exercise test) and the diaphragm, scalene muscles, sternocleidomastoid muscle, and rectus abdominis muscle (at rest) will be assessed with a muscle oxygen monitor.
Balance | Trough study completion, an average of 2 year
  Balance will be evaluated using a balance assessment device.
Balance (timed up and go test) | Trough study completion, an average of 2 year
  Balance will be evaluated a timed up and go test.
Physical activity level | Trough study completion, an average of 2 year
  A multi-sensor activity monitor will be used to assess the level of physical activity.

SECONDARY OUTCOMES:
Respiratory Muscle Strength | Trough study completion, an average of 2 year
  Maximal inspiratory and expiratory muscle strength will be evaluated using mouth pressure device.
Respiratory Muscle Endurance | Trough study completion, an average of 2 year
  The test will be started at 30% of maximum inspiratory pressure and the inspiratory threshold load will be increased by 10% of the maximal inspiratory pressure value every two minutes. New pressure loading will be maintained without removing the device from the mouth. If the individual cannot breathe 3 consecutive times, the test will be terminated by the physiotherapist. The total duration of the test and the maximum pressure value at which it continues to breathe for at least 1 minute will be multiplied. The value found will be recorded as the respiratory muscle endurance value.
Pulmonary function (Forced expiratory volume in the first second (FEV1)) | Trough study completion, an average of 2 year
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, forced expiratory volume in the first second (FEV1) will be evaluated.
Pulmonary function (Forced vital capacity (FVC)) | Trough study completion, an average of 2 year
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, forced vital capacity (FVC) will be evaluated.
Pulmonary function (FEV1/FVC) | Trough study completion, an average of 2 year
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, FEV1 / FVC will be evaluated.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | Trough study completion, an average of 2 year
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, flow rate 25-75% of forced expiratory volume (FEF 25-75%) will be evaluated.
Pulmonary function (Peak flow rate (PEF)) | Trough study completion, an average of 2 year
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, peak flow rate (PEF) will be evaluated.
Peripheral Muscle Strength | Trough study completion, an average of 2 year
  Shoulder abduction and knee extensor muscle strength using portable hand held dynamometer will be evaluated.
Trunk muscle endurance | Trough study completion, an average of 2 year
  Trunk muscle endurance will be evaluated with the pelvic bridge test and partial sit-up test.
Cough Strength | Trough study completion, an average of 2 year
  Cough strength will be assessed using a peak cough flow meter (PEFmeter) (ExpiRite Peak Flow Meter, China).
Dyspnea | Trough study completion, an average of 2 year
  Modified Borg Scale: The Modified Borg scale is a subjective scale that scores 0-10 for breathlessness and fatigue at rest and/or during activity. The lowest 0 points "not at all" the highest 10 points "very severe" means shortness of breath.
  The Modified Medical Research Council (MMRC) dyspnea scale will be used to determine the perception of dyspnea during activities of daily living.
Fatigue | Trough study completion, an average of 2 year
  Fatigue will be assessed with Fatigue Severity Scale (Turkish version). This scale includes 9 items and each item scores from 1 (strong disagreement) to 7 (strong agreement) point. Fatigue Severity Scale total score is calculates by deriving an arithmetic mean. Cut-score of over 4 means significant fatigue and higher score indicates more severe fatigue.
Disease Specific Quality of Life | Trough study completion, an average of 2 year
  Quality of life will be measured using Turkish version of European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 version 3.0 (EORTCQLQ). The cancer-specific questionnaire has 30 questions and incorporates five functional scales, three symptom scales, a global health status and several single items. All item scores are transformed to 0-100. Higher values indicate higher functional/health level in functional scales, a higher quality of life level in global health status and increased symptoms in symptom scales.

CONTACTS AND LOCATIONS:
Overall Officials: Gülsüm SERTTAŞ GÜVEN, MSc., Study Chair — Gazi University; Ece BAYTOK, MSc., Principal Investigator — Gazi University; Muhammet SAYAN, A. Prof. Dr, Principal Investigator — Gazi University; Ali ÇELİK, Prof. Dr., Principal Investigator — Gazi University; Meral BOŞNAK GÜÇLÜ, Prof. Dr., Study Director — Gazi University
Locations (1):
- Gazi University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooley ME. Symptoms in adults with lung cancer. A systematic research review. J Pain Symptom Manage. 2000 Feb;19(2):137-53. doi: 10.1016/s0885-3924(99)00150-5. PMID 10699541
- [Background] Miserocchi G, Beretta E, Rivolta I. Respiratory mechanics and fluid dynamics after lung resection surgery. Thorac Surg Clin. 2010 Aug;20(3):345-57. doi: 10.1016/j.thorsurg.2010.03.001. PMID 20619225
- [Background] Nomori H, Horio H, Fuyuno G, Kobayashi R, Yashima H. Respiratory muscle strength after lung resection with special reference to age and procedures of thoracotomy. Eur J Cardiothorac Surg. 1996;10(5):352-8. doi: 10.1016/s1010-7940(96)80094-7. PMID 8737692
- [Background] Granger CL, McDonald CF, Irving L, Clark RA, Gough K, Murnane A, Mileshkin L, Krishnasamy M, Denehy L. Low physical activity levels and functional decline in individuals with lung cancer. Lung Cancer. 2014 Feb;83(2):292-9. doi: 10.1016/j.lungcan.2013.11.014. Epub 2013 Nov 26. PMID 24360323
- [Background] Kocjan J, Gzik-Zroska B, Nowakowska-Lipiec K, Burkacki M, Suchon S, Michnik R, Czyzewski D, Adamek M. Thoracic surgery may alter body static balance via diaphragm dysfunction. PLoS One. 2022 Aug 31;17(8):e0273641. doi: 10.1371/journal.pone.0273641. eCollection 2022. PMID 36044444
- [Background] de Oliveira Vacchi C, Martha BA, Macagnan FE. Effect of inspiratory muscle training associated or not to physical rehabilitation in preoperative anatomic pulmonary resection: a systematic review and meta-analysis. Support Care Cancer. 2022 Feb;30(2):1079-1092. doi: 10.1007/s00520-021-06467-4. Epub 2021 Aug 21. PMID 34417883